





# INFORMACIÓN AL PARTICIPANTE Y CONSENTIMIENTO DE PARTICIPACIÓN

TITULO DEL ESTUDIO: "EVALUACIÓN DE LA EFICACIA DE LA N-ACETILCISTEÍNA PARA REDUCIR EL CRAVING Y PROLONGAR LA ABSTINENCIA DE PASTA BASE DE COCAÍNA"

Investigadora Responsable Investigador Alterno

: Carmen G. Betancur Moreno. Médico Psiquiatra. Benjamín Vicente Parada. Médico Psiguiatra. Carolina Gómez Gaete. Químico Farmacéutico.

María Paz Casanova Laudien, Estadística

Entidad Patrocinadora

Co-Investigadoras

Universidad de Concepción Financiado Por

: Fondo Nacional de Investigación y Desarrollo en Salud (FONIS)



#### INTRODUCCIÓN

A usted se le está invitando a participar en este estudio médico adjudicado en un concurso nacional de proyectos de investigación y desarrollo en salud (FONIS). Esta invitación se da en razón de ser usted paciente. Antes de decidir si participa o no, debe conocer y comprender cada uno de los siguientes apartados. Este proceso se conoce como consentimiento informado. Siéntase con absoluta libertad para preguntar sobre cualquier aspecto que le ayude a aclarar sus dudas al respecto. Una vez que haya comprendido el estudio y si usted desea participar, de manera libre y voluntaria, entonces se le pedirá que firme la hoja de Consentimiento Informado, adjunta al final de este documento, de la cual se le entregará una copia firmada y fechada.

#### 1. JUSTIFICACIÓN DEL ESTUDIO

Es necesario contar con un fármaco que nos permita ayudar a nuestros pacientes a disminuir y, en lo posible, a anular completamente el deseo (también conocido como "craving") de consumir pasta base de cocaína. A lo largo de los últimos años se han probado distintos fármacos para disminuir el craving de cocaína, pero no hay estudios realizados con fármacos que disminuyan este deseo de consumir pasta base (PBC). Es por eso que hemos elegido un fármaco que ya ha demostrado beneficios en la reducción del deseo de consumir cocaína, para evaluar la reducción del mismo síntoma en nuestros pacientes usuarios de pasta base. Este fármaco es la N- Acetilcisteína (NAC).

#### 2. OBJETIVO DEL ESTUDIO

A usted se le está invitando a participar en un estudio que tiene como objetivo evaluar el efecto de la NAC sobre el craving de PBC y la duración de la abstinencia de la misma, en pacientes con trastorno por consumo de esta sustancia.

#### 3. CENTROS DONDE SE REALIZARÁ EL ESTUDIO

El estudio se realizará en los siguientes centros de atención ambulatoria de la provincia de Concepción: COSAM de Lota, CentroTerapéutico Anun de Coronel, COSAM de Concepción y Servicio de Psiquiatría del Hospital Guillermo Grant

# 4. RAZÓN POR LA CUAL SE LE INVITA A PARTICIPAR

A usted se le invita a ser parte de este estudio ya que es paciente de uno de los centros elegidos para realizarlo y cumple con todos los criterios para ingresar al mismo.

#### 5. ACCESO A TRATAMIENTOS

Su participación en este estudio no implica en ningún caso que usted abandone o pierda la posibilidad de recibir el tratamiento estándar por el equipo de profesionales del COSAM o Centro de Salud donde estemos realizando nuestra investigación, si no, por el contrario, el protocolo de este estudio contempla que usted participe de él mientras se encuentra en el período de evaluación por el equipo de trabajo que normalmente le atendería en dicho centro. Ello implica que si ese equipo le indica, como parte de su proceso de evaluación previo a ingresar a tratamiento con ellos, que usted debe asistir a entrevista con psicólogo(a), asistente social u otro profesional que allí trabaje, así como a talleres psico-educativos, desayunos u otras intervenciones iniciales del centro, usted puede asistir a ellas tal y como lo hubiese hecho si no participase de este estudio.

Por otra parte, si los fármacos que nosotros le daremos como parte del estudio, no le aliviasen sus molestias principales, usted puede solicitar al médico del COSAM o Centro de Salud donde estemos realizando nuestra investigación, otro tipo de ayuda farmacológica (la cual se encuentra estadarizada según nuestro protocoo) y si dicho médico considerase que usted requiere de alguna otra medicación o intervención, puede indicarle que se retire de nuestro estudio cuando lo estime conveniente.

#### 5. DESCRIPCIÓN DEL ESTUDIO

En caso de aceptar participar en él, se le realizarán algunas preguntas sobre usted, sus hábitos de consumo de sustancias, sus antecedentes médicos y psiquiátricos, además de preguntas sobre las reacciones adversas que pudiera presentar con los fármacos utilizados, el deseo de consumo (o craving) de PBC y el tiempo sin uso de esta sustancia durante el estudio.

Versión 3. Fecha: 27-Abril-2017.

Investigadora Responsable: Dra. Carmen Gloria Betancur Moreno.

| <b>FOLIO</b> |
|--------------|

#### Este estudio consta de las siguientes fases:

- a. Evaluación médico-psiquiátrica: realizada por un médico psiquiatra, en la que se revisará su estado de salud general y salud mental (aplicando cuestionarios). Como parte de esta misma etapa de evaluación usted deberá realizarse un test de drogas en orina y exámenes bioquímicos generales (a través de una muestra de sangre de 10 cc= 2 cdtas. de té).
- b. Tratamiento: se le indicará un tratamiento farmacológico al azar, el cual puede ser 2 cápsulas cada 12 horas (2400 mg/día) de N-Acetilcisteína (NAC) ó 2 cápsulas cada 12 horas (2400 mg/día) de un compuesto farmacológicamente inactivo, por un período de cuatro semanas.
- c. Seguimiento: mientras se encuentre en tratamiento farmacológico, usted deberá asistir a controles dos veces por semana al centro de salud donde se está realizando el estudio. En estos controles se evaluará su evolución clínica, posibles efectos adversos por los fármacos, se le solicitará contestar algunos cuestionarios y se le tomarán tests de drogas en orina semanalmente.

#### 6. NÚMERO DE PACIENTES PARTICIPANTES DEL ESTUDIO

Para poder llevar a cabo de forma completa este estudio, será necesario contar con 106 (ciento seis) pagiéntes, mayores de 18 años de edad y de ambos sexos, que participen de él.

#### 7. DURACIÓN ESPERADA:

a. Del estudio: 2 (dos) años.

b. De su participación: 4 (cuatro) semanas.

## 8. BENEFICOS DERIVADOS DE SU PARTICIPACIÓN

Al ser éste un estudio en el cual se evalúa el efecto de un fármaco sobre los síntomas de abstinencia de PBC, usted podría beneficiarse logrando reducir sus ansias (o *craving*) por consumir PBC y prolongar sus días sin usar esta droga, lo que no podemos garantizarle actualmente. Por otra parte, los resultados obtenidos de este estudio permitirán ayudar al conocimiento médico sobre este tema.

## 9. RIESGOS DERIVADOS DE SU PARTICPACIÓN

La N-Acetilcisteína (NAC) es un fármaco utilizado en Chile desde hace varios años y autorizado por el Instituto de Salud Pública (ISP) para la protección de la función renal en los pacientes sometidos a exámenes con medio de contraste, para facilitar la eliminación del paracetamol en casos de intoxicación por dicho fármaco y para facilitar la eliminación de secreciones (mucolítico) en pacientes con cuadros respiratorios como bronquitis o fibrosis quística.

Algunos efectos colaterales que pudiese presentar por el uso de este fármaco son: prurito y/o rash cutáneo (picazón o manchas rojas en la piel), cefalea (o dolor de cabeza), flatulencia y/o diarrea, acumulación de secreciones bronquiales, leve aumento de la presión arterial, sudoración y leve aumento del apetito. Todos ellos son efectos leves y manejables.

#### 10. MODALIDAD DE COMUNICACIÓN DE EVENTOS ADVERSOS

A usted se le preguntará, en las respectivas entrevistas de evaluación y seguimiento, acerca de los posibles eventos adversos relacionados con el uso de la medicación indicada según el protocolo de estudio. Sus respuestas serán registradas en una ficha clínica estandarizada, creada especialmente para este estudio. Además usted podrá informar directamente al equipo investigador, a través del teléfono y/o el correo indicado más abajo, acerca de alguna reacción adversa que a usted le preocupe o que a su juicio (o el de un clínico) requiera de atención médica.

En caso de que usted reporte algún evento adverso relacionado con la medicación indicada, éste será notificado al Instituto de Salud Pública de Chile (ISP) a través de un formulario estándar, además de reportarlo previamente al Comité de Farmaco-Vigilancia correspondiente y al Comité Ético Científico del Servicio de Salud Concepciónse, junto con otorgarle la ayuda médica que usted requiera cuando informe del evento, cuyo costo no será asumido por ud. en ningún caso.

## 11. RESPONSABILIDADES DEL PARTICIPANTE/PACIENTE

Su decisión de participar en este estudio es completamente libre y voluntaria. No habrá ninguna consecuencia desfavorable para usted, en caso de no aceptar la invitación a participar en él. Los controles para fines del estudio se realizarán en las mismas visitas planeadas por el equipo clínico del centro de salud como parte del proceso de evaluación y tratamiento inicial habitual, por lo cual usted no tendrá que hacer gasto alguno durante el estudio. Tampoco recibirá pago por su participación.

# 12. TÉRMINO ANTICIPADO

Por otra parte, si usted decide participar en este estudio, puede retirarse en el momento que lo desee, aún cuando el investigador responsable no se lo solicite, pudiendo informar o no, las razones de su decisión, la cual será respetada en su integridad.

# 13. CONFIDENCIALIDAD DE LA INFORMACIÓN

Toda la información que se recoja en este estudio será confidencial y no se usará para ningún otro propósito que no sean los de ésta. Así también se garantiza la privacidad de las opiniones y juicios emitidos por usted. Toda la información obtenida será custodiada por la Investigadora Responsable.

| FOLIO |
|-------|

## 14. COMUNICACIÓN DE LOS RESULTADOS

Los resultados del tratamiento de cada sujeto participante del estudio serán entregados directamente a él(ella) al finalizar el estudio. Además los resultados globales del mismo serán comunicados tanto a la entidad patrocinadora (Universidad de Concepción) como a quien financia el estudio (FONIS) a través de informes escritos que serán enviados directamente a estas entidades, resguardando la confidencialidad de la información de sus participantes. Por otra parte, los resultados de este estudio serán comunicados a la comunidad científica nacional e internacional, a través de publicaciones en revistas debidamente acreditadas para ello, con el mismo resguardo previamente mencionado.

### 15. CONTACTO PARA EMERGENCIAS / CONTACTO CON COMITÉS DE ÉTICA

Si usted tiene alguna emergencia derivada de este estudio o requiere información adicional sobre su participación durante cualquier etapa del mismo, puede comunicarse con la Investigadora Responsable, Dra. Carmen Gloria Betancur Moreno, a los teléfonos 41-2212006 ó +56(9)930276194 o al correo fonisnac@udec.cl. De no recibir respuesta puede contactarse con el Dr. José Becerra, Presidente del Comité de Ética de la Universidad de Concepción, al teléfono (41) 2204302 o con la Dra. María Antonia Bidegain S., Presidente del Comité Ético Científico del Servicio de Salud Concepción, ubicado en San Martín 1436, al teléfono (41) 2722745.

Si considera que no hay dudas ni preguntas acerca de su participación, puede, si así lo desea, firmar la Declaración de Consentimiento Informado que forma parte de este documento.

# DECLARACIÓN DE CONSENTIMIENTO INFORMADO Título del estudio: "Evaluación De La Eficacia De La N-Acetilcisteína Para Reducir El Craving Y Prolongar La Abstinencia De Pasta Base De Cocaína" he leído y comprendido la información anterior y mis preguntas han sido respondidas de manera satisfactoria. He sido informado y entiendo que los datos obtenidos en el estudio pueden ser publicados o difundidos con fines científicos. Consiento voluntariamente en participar de este estudio de investigación, entendiendo que puedo retirarme en cualquier momento de él sin recibir sanción alguna por ello. Recibiré una copia firmada y fechada de esta hoja de consentimiento y, al firmarlo, sé que no renuncio a ninguno de mis derechos legales como paciente. Firma del Participante/Paciente Fecha Esta parte debe ser completada por el Investigador Responsable: He explicado al Sr(a). la naturaleza y los propósitos de la investigación; le he explicado acerca de los riesgos y beneficios que implica su participación. He contestado a las preguntas a satisfacción del Participante/Paciente y he preguntado si tiene alguna duda. Una vez concluida la sesión de preguntas y respuestas, se procedió a firmar el presente documento. Nombre y Firma del(la) Investigador(a) Responsable Fecha Nombre y Firma del(la) Director(a) o Delegado(a) del Centro de Salud DECLARACIÓN DE REVOCACIÓN DEL CONSENTIMIENTO Título del estudio: "Evaluación De La Eficacia De La N-Acetilcisteína Para Reducir El Craving Y Prolongar La Abstinencia De Pasta Base De Cocaína" Investigadora Responsable: Carmen Gloria Betancur Moreno. Médico Psiquiatra. Nombre del paciente: \_\_ \_\_ RUT: \_\_\_\_ Firma del Participante/ Paciente Fecha Testigo Fecha

Versión 3. Fecha: 27-Abril-2017.

Investigadora Responsable: Dra. Carmen Gloria Betancur Moreno.

Nombre y Firma del(la) Investigador(a) Responsable

Fecha